CLINICAL TRIAL: NCT06789419
Title: Predicting Epileptogenic Tubers in Patients with Tuberous Sclerosis Complex Using a Fusion Model Integrating Lesion Network Mapping and Machine Learning
Brief Title: Predicting Epileptogenic Tubers in Patients with Tuberous Sclerosis Complex
Status: Completed | Type: Observational
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Shuli Liang, Director, Beijing Children's Hospital
Other Study IDs: TSC-MRI
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2023-06

CONDITIONS: Tuberous Sclerosis Complex
Keywords: TSC; TSC MRI
MeSH Terms: conditions — Tuberous Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TSC: TSC

SUMMARY:
Accurate localization of epileptogenic tubers (ETs) in patients with tuberous sclerosis complex (TSC) is essential but challenging because ETs lack distinct pathological or genetic markers that differentiate them from other cortical tubers. Approximately 60% of patients fail to have their ETs identified through noninvasive preoperative evaluations, highlighting the clinical need for an efficient, noninvasive ET localization method.

Using MRI data from training datasets, we developed a novel noninvasive fusion model that combines a risk model based on lesion network mapping with a prediction model using brain functional connectivity and random forest algorithms. A retrospective analysis was conducted on TSC patients with epilepsy who underwent resective surgery. Tubers were classified as true-ETs, false-ETs, or true non-ETs based on resection locations and postoperative seizure-freedom. The model calculated and ranked the ET probability for each tuber for every patient, and its accuracy was assessed based on postoperative seizure outcomes.

ELIGIBILITY:
Inclusion Criteria:

(1) male or female patients aged ≥6 months; (2) patients meeting the diagnostic criteria for TSC according to Northrup's guidelines;17 (3) patients in whom the clinical evaluation determined that a single surgical target, or hypothesized primary EZ, was identified by a multidisciplinary specialist team at epilepsy centers of Beijing Children's Hospital, PLA General Hospital, or Shenzhen Children's Hospital in China; (4) patients who underwent resective surgery between July 2016 and June 2023, with a 1-year follow-up completed by June 2024; and (5) availability of patients with available preoperative and postoperative MRI T2-Flair imaging.

Exclusion Criteria:

* (1) patients with a history of craniotomy, serious head injury, neuromodulation therapy, or corpus callosotomy before or within one year after the resective surgery; and (2) subjects lacking key clinical or MRI data. This study was approved by the Ethics Commission of Beijing Children's Hospital.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
seizure freedom after surgery | From enrollment to the end of treatment at 1 year

IPD SHARING:
Plan to Share IPD: No